CLINICAL TRIAL: NCT02408601
Title: A Clinical Trial to Assess the Retention and Caries Preventive Effect of Resin Based Sealants Versus ART Sealants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr. Praveen B.H (Other)
Collaborators: Kamineni Institute of Dental Sciences (Other)
Responsible Party: Sponsor-Investigator, Dr. Praveen B.H, A randomized controlled clinical trial to assess the retention and caries preventive effect of Resin based sealant versus ART sealant among the 6-12 yr old school children of a district in India. A 24 months follow up study., Kamineni Institute of Dental Sciences
Organization: Kamineni Institute of Dental Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KamineniIDS
Record Dates: First submitted 2015-03-24; First posted 2015-04-03 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): split mouth study. one side of the arch that is the lower left permanent 1st molar will be receiving resin based sealants.
  Application of the resin sealants as per the standard instructions of the manufacturer
  Helioseal -F ( Resin based sealant)
  1. isolate the tooth surface
  2. etch the fissure anatomy with 37% phosphoric acid for 20 seconds
  3. wash the tooth surface and dry it. No salivary contamination is accepted
  4. using a syringe based system, apply the sealant onto the fissures, do not overfill the fissures, run an explorer along the fissures to avoid any air entrapment.
  5. light cure the sealant
  6. check for high points and the occlusion
  Interventions: Other: Helioseal - F
- Group 2 (Experimental): split mouth study. one side of the arch that is the lower right permanent 1st molar will be receiving ART sealants.
  Application of the ART sealants as per the standard instructions of the manufacturer
  1. isolate the tooth surface
  2. condition the fissure anatomy using a GC conditioner for 10 seconds
  3. wash the conditioner by using a cotton pellet for a couple of times, do not use a three way syringe.
  4. dry the tooth surface
  5. mix the GIC according to the standard powder: liquid ratio
  6. place the mix onto the fissures using a plastic spatula
  7. apply pressure on the occlusal surface with a gloved index finger( the gloved index finger must be coated with petroleum jelly)
  8. apply pressure for 10-15 sec and withdraw the finger in a sideways motion
  9. scrap out the excess material
  10. check for the high points and the occlusion
  11. apply petroleum jelly onto the GIC mix
  12. advice patient not to eat or drink for 30 minutes.
  Interventions: Other: ART sealant

INTERVENTIONS:
Other: Helioseal - F — Helioseal -F ( Resin based sealant)
  1. isolate the tooth surface
  2. etch the fissure anatomy with 37% phosphoric acid for 20 seconds
  3. wash the tooth surface and dry it. No salivary contamination is accepeted
  4. using a syringe based system, apply the sealant onto the fissures, do not overfill the fissures, run an explorer along the fissures to avoid any air entrapment.
  5. light cure the sealant
  6. check for high points and the occlusion
  Arms: Group 1
Other: ART sealant — Fuji IX extra strength
  1. isolate the tooth surface
  2. condition the fissure anatomy using a GC conditioner for 10 seconds
  3. wash the conditioner by using a cotton pellet for a couple of times, do not use a three way syringe.
  4. dry the tooth surface
  5. mix the GIC according to the standard powder: liquid ratio
  6. place the mix onto the fissures using a plastic spatula
  7. apply pressure on the occlusal surface with a gloved index finger( the gloved index finger must be coated with petroleum jelly)
  8. apply pressure for 10-15 sec and withdraw the finger in a sideways motion
  9. scrap out the excess material
  10. check for the high points and the occlusion
  11. apply petroleum jelly onto the GIC mix
  12. advice patient not to eat or drink for 30 minutes.
  Arms: Group 2

SUMMARY:
Background and study aims:

The investigators are carrying out a clinical trial of two different sealant materials to compare the retentivity and decay inhibiting properties of the above said materials. it is a split mouth study, wherein the 2 sealant materials will be placed on the exactly opposite placed molars of 198 healthy school children in the age group between 6 - 12 yrs of age.

who can participate? school children in the age group between 6 - 12 yrs of age with non decayed contra lateral permanent 1st molars at a school in the southern part of India.

what does the study involve? over a period of 24 months, the retentivity and the decay preventing effects of these two sealant materials( RESIN BASED SEALANTS AND ART SEALANTS) will be clinically assessed by us.

possible benefits/ risks of participating in the trial the participants will be not be exposed to any kind of risks as it is a non invasive procedure the possible benefits may be preventing decay to the permanent molar in the long run

study start date/duration of the study? MARCH 2015 is the month wherein the sealant applications have started and expected to last till the April of 2017

funding? self funded study

DETAILED DESCRIPTION:
Pits and fissures in the first molars are the most susceptible sites for dental caries in the permanent dentition and contemporary studies show specifically that 85% or more of the caries is nested in the above-mentioned sites . Thus, prevention of caries in these tooth sites is of crucial importance in keeping a sound permanent dentition.

Sealing the pits and fissures of molars and premolars for prevention of dental caries was first introduced in the 1960s . It is now accepted as a highly effective method in preventing dental caries .

Prominently, there are basically two types of sealant materials..i.e resin based sealants which are flowable composite resins and Glass ionomer based sealants. Reading through the literature, it is well understood that the resin based sealants are more retentive than the GIC based sealants mainly because the enamel surface is etched prior to the placement and it is dispensed through syringes, thereby it generally adapts well to the surfaces. GIC sealants are known to be equally effective when to comes to caries prevention, but generally are far less retentive than the resin based sealants. the main issue regarding the placement of resin based sealants is that it is a cumbersome procedure requiring strict isolation. Looking at a dental public health point of view, especially in a country like India, the use of resin based sealants at outreach centres will be a problem because of the lack of adequate infrastructure.

To counter the limited applicability of resin based sealants in a field setting, the use of a high viscosity GIC sealant is advocated here. The high viscosity GIC sealant has a better compressive strength to take on the occlusal stress and thereby it is expected that the retention of the ART sealant (High viscous GIC sealant) using the ART technique (finger press technique) would be better than the conventional GIC based sealants. Till date, a very limited number of studies have been performed on the comparison between the ART sealant and the resin based sealant( gold standard) and thereby, this study has been conceived to assess the retentivity and the caries preventive effect of the above two systems.

The null hypothesis states that there is no expected difference between resin based sealants and ART sealants

Based on the statistical analysis, the sample size for this study has been estimated to be 198 subjects. ethical clearance has been obtained from the IRB of the dental school and informed consent obtained from all the participating subjects. This is a spilt mouth study, wherein on side, resin based sealants are placed and on the other side, the ART sealants are placed. All the participating 198 subjects do have a caries free lower permanent lower 1st right and left molars.

The sealants are placed according to the manufacturer s instructions. after placements, the retention and the caries preventive effects are followed up progressively for a period of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* children belonging to high caries risk group
* 1st permanent molars with an exaggerated pit and fissure system

Exclusion Criteria:

* non cooperative children excluded
* children with history of systemic diseases
* parents haven't given their consent for this preventive therapy

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2015-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
retention rate as given by the simonsons criteria | 24 months

SECONDARY OUTCOMES:
caries incidence | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Haricharan Bhoopathi, M.D.S, Principal Investigator — Kamineni Institute of Dental Sciences
Locations (1):
- Divya Bala School, Bhongir, Andhra Pradesh, India